CLINICAL TRIAL: NCT05846932
Title: Preliminary Efficacy of Occupational Therapy Integrating Horses on Self-regulation in Youth With Autism Spectrum Disorder
Brief Title: Preliminary Efficacy of Occupational Therapy Integrating Horses on Self-regulation in Youth With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4049; 1R21HD109957-01 (NIH)
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: occupational therapy; hippotherapy; equine-assisted services; self-regulation
MeSH Terms: conditions — Autism Spectrum Disorder; Self-Control

STUDY DESIGN:
Intervention Model Description: Youth with be randomized to either receive occupational therapy integrating horses (OTEE HORS) or occupational therapy in a clinic (OT Clinic)
Who Masked: Outcomes Assessor
Masking Description: The research assistant that rates goal attainment at the conclusion of therapy will be asked to participants' intervention assignment (OTEE HORS v OT Clinic).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational Therapy Integrating Horses (Experimental): 10 weeks of occupational therapy focused on self-regulation skills, provided while participants are riding horses
  Interventions: Behavioral: OTEE HORS
- Occupational Therapy in a Clinic (Active Comparator): 10 weeks of occupational therapy focused on self-regulation skills, provided in a traditional clinic environment
  Interventions: Behavioral: OT Clinic

INTERVENTIONS:
Behavioral: OTEE HORS — 10 weeks of occupational therapy focused on teaching and practicing self-regulation skills, provided while participants are riding horses
  Arms: Occupational Therapy Integrating Horses
Behavioral: OT Clinic — 10 weeks of occupational therapy focused on teaching and practicing self-regulation skills, provided in a traditional clinic
  Arms: Occupational Therapy in a Clinic

SUMMARY:
The goal of this clinical trial is to learn about occupational therapy integrating horses for autistic youth. The main questions it aims to answer are:

* Does occupational therapy integrating horses improve self-regulation in autistic youth
* Does occupational therapy integrating horses affect salivary cortisol and alpha-amylase

Participants will receive 10 weeks of occupational therapy, and will be asked to provide saliva samples each week.

Researchers will compare occupational therapy integrating horses to occupational therapy in a clinic to see if integrating horses affects self-regulation.

DETAILED DESCRIPTION:
The goal of this project is to quantify the unique benefits of integrating horses in occupational therapy compared to occupational therapy in a clinic (i.e., OTEE HORS vs. OT Clinic) for improving self-regulation in youth with ASD.

To address both aims we will randomize 64 youth with ASD ages 6-11 years old to OTEE HORS or OT clinic.

Specific Aim 1: Examine the preliminary efficacy of OTEE HORS compared to OT Clinic on self-regulation. Hypotheses: The OTEE HORS group will demonstrate significantly larger improvements than the OT Clinic group in five domains of self-regulation (hyperactivity [primary], irritability, emotional reactivity, dysphoria, and individual goal attainment).

Specific Aim 2: Identify potential physiological mechanisms that explain how integration of horses in occupational therapy impacts self-regulation in youth with ASD. Hypotheses 2A & B: The OTEE HORS group will demonstrate significantly larger decreases in salivary cortisol after each 60-minute therapy session and after the 10-week treatment course in comparison to the OT Clinic group. Hypotheses 2C & 2D: The OTEE HORS group will demonstrate significantly greater increases in salivary alpha-amylase after each 60-minute therapy session, and significantly greater decreases in salivary alpha-amylase over time as measured after the 10-week treatment course in comparison to the OT Clinic group. Exploratory Hypothesis 2E: Changes in physiological measures will significantly correlate with changes in Aim 1 behavioral measures.

ELIGIBILITY:
Inclusion Criteria:

* meet clinical cut-offs for ASD on the Autism Diagnostic Observation Schedule, Second Edition(ADOS-2) and Social Communication Questionnaire (≥ 11)
* nonverbal IQ≥65 on Leiter International Performance Scale Third Edition (Leiter-3)
* verbally fluent defined by meeting standard administration criteria for ADOS-2 module 3
* score >10 on the irritability subscale of the aberrant behavior checklist
* able to tolerate a helmet and ride a horse for 10 minutes while following safety rules
* and able to provide a saliva sample

Exclusion Criteria:

* weigh more than 200 pounds
* smoke or regularly use steroids
* receive outpatient occupational therapy
* have 10+ hours horseback riding experience in the previous 6 months
* history of animal abuse or phobia of horses
* have a sibling previously enrolled in the study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist, Community | Week 1 & Week 10
  Parent-report checklist of problematic behaviors related to hyperactivity and irritability

SECONDARY OUTCOMES:
Change in Emotional Dysregulation Inventory | Week 1 & Week 10
  Parent-report measure of emotional reactivity and dysphoria
Change in Concentration of Salivary Cortisol | Week 1, Week 6, Week 10
Change in Concentration of Salivary Alpha-amylase | Week 1, Week 6, Week 10
Goal Attainment using Goal Attainment Scale | Week 10
  Attainment of individualized self-regulation goals. Goal attainment scales range from -2 to +2 where higher values indicate greater progress towards individual goal.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany C Peters, PhD, Principal Investigator — Colorado State University
Locations (1):
- Temple Grandin Equine Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in an appropriate data repository, such as the "Data and Specimen Hub" (DASH) or the "National Database for Autism Research" (NDAR). Data will be shared no later than the acceptance for publication of the main findings from the final dataset. Salimetrics will discard saliva samples after testing, and therefore saliva samples will not be available for sharing.
Supporting Information: ICF
Time Frame: We will share in an appropriate data repository indefinitely, no later than the acceptance for publication of the main findings from the final dataset

REFERENCES:
- See also: Temple Grandin Equine Center Denver — https://csuspur.org/tgec/

DOCUMENTS (1):
  • Informed Consent Form (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT05846932/ICF_001.pdf